CLINICAL TRIAL: NCT06005623
Title: Impact of Motivational Feedback on Levels of Physical Activity and Quality of Life by Activity Monitoring Following Knee Arthroplasty Surgery - Randomized Controlled Trial Nested in a Prospective Cohort (KneeActivity)
Brief Title: Motivational Feedback Following Total or Unicompartmental Knee Arthroplasty
Acronym: KneeActivity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Gigtforeningen (Other); Region of Southern Denmark (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, Anders Holsgaard Larsen, Professor, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OUH KneeActivity
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Knee Arthropathy
Keywords: Physical activity; Motivational Feedback; Rehabilitation; Tele-Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Multicenter randomized (1:1) parallel-group intervention study with blinded statistical analysis towards group allocation. Patients will be randomized to activity tracking and motivational feed-back by gamification for patient self-mobilization (INT) or 'care-as-usual' including activity tracking without motivational feed-back (CON).
Who Masked: Investigator
Masking Description: Data will be analyzed by the PhD student blinded towards group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Activity tracking and motivational feed-back by gamification.
  Interventions: Device: SENS Motion + Motivational Feedback
- Care as usual (No Intervention): Activity tracking without motivational feed-back

INTERVENTIONS:
Device: SENS Motion + Motivational Feedback — To weeks prior to surgery and in a 12-week period following discharge after TKA/UKA patients will be equipped with a discrete patch and built-in accelerometer (SENS Motion, Denmark, Copenhagen) attached on the thigh of the leg not undergoing surgery.
  Following discharge after TKA/UKA patients randomized to the intervention-group will receive the app ("SENS motion"). On their provided app, patients will be able to choose between two tabs. Tab 1 will allow patients to view predefined goals, all of which are locations in a self-selected city. The sensor will measure the physical activity and daily rhythm of the patient, and accelerometer counts will be converted into daily steps, which will be visible to the patients. In Tab 2, patients will be able to see graphical representations of their daily activity as well as their history during the period in which they have worn the accelerometer. The graphical representations include: Daily steps, physical active minutes, and type of activity.
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial (RCT) nested in a prospective cohort study is to investigate whether physical activity (PA) following total knee arthroplasty (TKA) or unicompartmental knee arthroplasty (UKA) can be optimized by the use of an activity tracking device including motivational feedback in comparison with activity tracking without feedback. Furthermore, the project will investigate the predictive value of PA level prior to TKA/UKA for the length of stay, return to work, and quality of life.

The main hypothese of the study are:

RCT study:

* Using an activity tracking device, including motivational feed-back on PA show a superior short-term effect on increased PA (Total counts; primary outcome measure), physical functioning, return to work, and quality of life in comparison with no motivational feed-back from the activity tracker, defined as 'care as usual', in TKA and UKA patients
* Using an activity tracking device, including motivational feedback, will have a superior effect on step counts, activity types and pain compared to the standard care, in TKA and UKA patients

Prospective cohort:

* PA prior to TKA or UKA can work as a predictive measure for function and quality of life following surgery
* PA prior to TKA or UKA can work as a predictive measure for the length of hospital stay and return to work

Patients will be randomized to activity tracking and motivational feed-back by gamification for patient self-mobilization (Intervention-group) or 'care-as-usual' including activity tracking without motivational feed-back (Control-group). Patients not eligible and/or willing to participate in the RCT study, will be offered to participate in a prospective non-interventional cohort study.

DETAILED DESCRIPTION:
Background:

Worldwide over a million patients receive a TKA or UKA each year and in Denmark more than 10,000 TKA and UKA's are performed annually, and the lifetime risk of symptomatic osteoarthritis (OA) of the knees are 45%. Despite being considered a successful intervention, 15-25% of patients following TKA are not satisfied with their output, which to some degree may be associated with reduced daily physical activity (PA). Few scientific studies have examined how daily PA is affected by TKA and how it might affect rehabilitation. It is unknown if a focus on increased PA in everyday life after return from hospital might improve rehabilitation and patient satisfaction. The current study addresses this 'gap' in science with high-level clinical evidence, to investigate if a novel technology on motivational feed-back regarding PA can be introduced to assist patients with a better rehabilitation following TKA or UKA.

Aim:

The aim of this randomized controlled trial (RCT) nested in a prospective cohort is to investigate whether PA following TKA or UKA can be optimized by the use of an activity tracking device including motivational feedback in comparison with activity tracking without feedback. Furthermore, a prospective cohort will investigate the predictive value of PA level prior to TKA/UKA for the post-surgical length of stay, return to work, and quality of life.

Trial design overview:

Design:

Randomized, blinded, two-arm, multi center trial. 150 patients scheduled for TKA or UKA will be recruited through Odense University Hospital (Svendborg and Odense) and Vejle Hospital. Patients will be randomized to 12 weeks of activity tracking and motivational feed-back by gamification for patient self-mobilization (Intervention group) or 'care-as-usual' including activity tracking without motivational feed-back (control group).

Patients that are not eligible and/or willing to participate in the RCT study will be offered to participate in a prospective non-interventional cohort study where the main outcome are self-reported disability, generel health, return to work, pain medication, overall experience with TKA or UKA.

SENS Motion:

SENS Motion (SENS Innovation ApS, Copenhagen, Denmark) is a wireless medical accelerometer for collecting objectively PA data. SENS Motion has developed a patient app with gamification/motivational feed-back to enhance PA. SENS Motion is CE marked as a medical device. SENS Motion has no right to unpublished study data and is neither financially nor personally involved in this trial. None in the study group is related to SENS Motion.

Blinding:

The primary investigator will be blinded to allocation and will not participate in randomization of patients. The statistical analysis will be performed on allocation codes only and thus the data analysts will be blinded in relation to intervention allocation. Blinding to intervention of patients, surgeon, and nurses (healthcare providers) will not be possible due to the nature of the intervention.

Randomizing and database:

Randomization is performed internet-based using REDCap Randomize, allocated 1:1. The randomization itself takes place right after the surgery. The randomization is performed as a block randomization in blocks of 2, 4 and 6. No stratifications are applied to the randomization, and the primary investigator is blinded regarding the permuted blocking strategy. A data manager, with no clinical involvement in the trial, prepares the randomization sequence. The allocation is concealed in a password-protected computer file.

Compliance:

Patients in the control group will have the app installed on their smartphones without motivational feedback, solely for transferring data from the activity tracker. To prevent data loss, weekly SMS messages will remind both intervention and control groups to open their SENS app during the week. No standard for adherence in app interventions has been established previously. The implementation aims for a 70% adherence rate, indicating that the intervention group will interact with the app and obtain motivational feedback for 5 out of 7 days weekly.

All patients will receive written information on how to attach the sensor, use the app (without a tablet), and use the tablet with motivational feedback. Moreover, all patients will receive a link to a YouTube video presenting the project and providing instructions on how to use the equipment.

Time points Assessment will be performed at baseline two weeks prior to surgery and randomization, following the intervention (14 weeks post baseline) (the primary endpoint) and a long term follow-up at 12 months post baseline.

Sample size:

Sample size is estimated using total accelerometer counts per day from a previous publication on TKA patients. Between-group difference in change score of 50.500 activity counts per day representing ≈ 1/3 standard deviation and a change of ≈17% is considered clinically relevant. To achieve a statistical power of 80% (β=0.80), using a standard deviation of 101.000 counts per day pre- and post-intervention, and allowing the detection of statistically significant differences at an α level of 0.05 (two-tailed testing), a sample size of n = 62 is estimated for each group. Allowing for dropout a recruitment of 150 patients (in total) is planned.

Main comparative analyses between groups will be performed by using an intention-to-treat analysis. Between-group mean differences and 95% confidence intervals will be estimated with a general linear model in which the patients baseline score is entered as a covariate and adjusted for potential baseline differences (age, sex, BMI). In addition to the intention-to-treat analysis, a per-protocol analysis will be also be conducted.

Ethics:

The study has been submitted to the regional Committee for Medical Research Ethics, which has assessed the project as "not subject to notification", Project-ID: S-20222000 - 171. Finally, The Danish Medicines Agency has declared no need for further permission to carry out the study.

Qualitative study:

A qualitative study using iterations where patients and healthcare professionals through interviews provided input for improvements of the current technology was initiated to tailor the technological maturation of the SENS App for the current patient group. Evaluation and patient involvement will be based on interviews of ten patients. Feed-back from the focus group will be implemented in an updated app-version. The first iteration was in augus t2021, the second was in feburary 2023, the last iteration is planed in september 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40-85 years
2. patients scheduled for primary TKA or UKA
3. understanding both verbal and written Danish language.

Exclusion Criteria:

1. Difficulty adhering to the study protocol
2. Refusal of standard care
3. Known- or newly diagnosed malignancy or palliative care
4. Participation in an interventional clinical trial during the last 3 months potentially interacting with the aims of the current study.
5. Do not own a smartphone

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Between-group change score of total daily PA (accelerometer counts) | Baseline and 12 weeks
  PA will be evaluated by SENS Motion as described above. The primary outcome measure is the between-group change score of total daily PA (accelerometer counts) from baseline to 12 weeks following discharge. Accelerometer counts per day is a cumulative and validated variable based on raw accelerometer data in 3 planes and is a proxy for total daily PA

SECONDARY OUTCOMES:
Physical active minuts (Between-group change) | Baseline and 12 weeks
  Physical active minutes per day measured with SENS motion.
Physical activity (Between-group change) | Baseline, 12 weeks and 12 months
  Patient-reported physical activity will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF measures activity over the past week in four different intensity levels, including 1) vigorous activities, 2) moderate activities, 3) walking, and 4) sitting. Higher value equals higher level of activity.
Patient satisfaction and patient reported outcome measures (Between-group change) | Baseline, 12 weeks and 12 months
  The OKS (Oxford Knee Score) is a validated 12-item questionnaire evaluate outcomes following TKA. It was translated into Danish in 2009, its validity in Danish has not been confirmed. The questionnaire generates scores ranging from 0-48, with a score of 4 representing the best outcome post-TKA. Each item response is graded between 0-4. A Danish study found that the minimal important change is 8.
Quality of Life (Between-group change) | Baseline, 12 weeks and 12 months
  The EQ-5D-5L (European Quality of Life - 5 Dimensions) is a validated survey for measuring HRQoL It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The outcome is reported on a scale of 1-5 where 1 is no problems and 5 is extrem problems. The EQ-5D-5L is validated in knee OA patients referred for knee replacement surgery [43].
Return to work in day-surgery (Between-group change) | 12 weeks, 12 months
  For patients active in the labor market, time on sick leave before returning to work (full time or part time) will be assessed by a questionnaire.
Global Perceived Effect (GPE) (Between-group change) | 12 weeks, 12 months
  Global Perceives Effect questions will be used for measuring the participants' overall experience with the TKA or UKA. A 5-point likert scale using the following answers will be used "Much worse", "Little worse", "The same", "Little better", and "Much better.

OTHER OUTCOMES:
Activity types (Between-group change) | Baseline and 12 weeks
  Activity types evaluated by SENS motion i.e. time spent sleeping/resting, standing, walking, and cycling will be evaluated.
Post-OP pain (Between-group change) | 12 weeks
  The patients receive weekly text message (SMS) with a question about their knee-pain. They will be asked to rate their pain on a NRS scale from 0-10, where 0 corresponds to no pain and 10 correspoinds to worst imaginable pain.
Use of POST-op pain medication (Between-group change) | 12 weeks
  Patients will receive a SMS with a question about their use of pain medication the last week. The SMS have 3 options: 1. No use of pain medication, 2. non-prescription medicine (e.g. Panodil, Pamol, Ibumetin), and 3. strong-painkillers (e.g. Morphine, Tramadol).

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie D Skov, MD, Principal Investigator — Odense University Hospital and Institute of Clinical Research, SDU; Anders Holsgaard-Larsen, Professor, Study Director — Odense University Hospital and Institute of Clinical Research, SDU
Locations (4):
- Denmark (4):
  - Herlev Gentofte Hospital, Hellerup, Region Sjælland
  - Odense University Hospital, Odense
  - Odense University Hospital, Svendborg
  - Lillebaelt Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skov CD, Lindberg-Larsen M, Wiil UK, Varnum C, Schmal H, Jensen CM, Holsgaard-Larsen A. Impact of motivational feedback on levels of physical activity and quality of life by activity monitoring following knee arthroplasty surgery-protocol for a randomized controlled trial nested in a prospective cohort (Knee-Activity). BMC Musculoskelet Disord. 2024 Oct 2;25(1):778. doi: 10.1186/s12891-024-07878-0. PMID 39358699